CLINICAL TRIAL: NCT05728073
Title: Does Subtotal Cholecystectomy Rate for Acute Cholecystitis Change With a Previous ERCP?
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Turgut Donmez, Ass. Prof. Dr., Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 20230205
Record Dates: First submitted 2023-02-05; First posted 2023-02-14 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Cholecystectomy, Laparoscopic; Cholangiopancreatography, Endoscopic Retrograde
Keywords: Acute Cholecystitis, Laparoscopic Subtotal Cholecystectomy
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard (non-ERCP) Group: Patients who underwent surgery for acute cholecystitis without a previous ERCP history.
- ERCP group: Patients who underwent surgery for acute cholecystitis with a previous ERCP history.
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: ERCP — Patients separated to two groups according to having a ERCP history before the operation
  Groups: ERCP group

SUMMARY:
Study is designed to investigate whether the history of ERCP is associated with subtotal cholecystectomy rates in patients underwent laparoscopic cholecystectomy operations with the diagnosis of acute cholecystitis.

DETAILED DESCRIPTION:
The results of patients who underwent surgery for acute cholecystitis in a single center between January 2016 and December 2019 were included and evaluated retrospectively.

Primary outcome was subtotal cholecystectomy rate. Secondary outcomes were conversion to open, complications and serious complications. Within examining demographic findings, operative records (rates for subtotal cholecystectomy and conversion to open, operative duration) and follow-up results (postoperative complications, serious complications, length of hospital stay and mortality) for all cases were investigated. Complications that Clavien-Dindo Score ≥ 3 accepted as serious complication. Intraoperative detection of gallbladder perforation was also noted and included in comparison. Any biliary tract complication that needed any percutaneous or endoscopic intervention to handle was named as "biliary leak" in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated with the diagnosis of acute cholecystitis with an age greater or equal to 18 years old in a single center between January 2016 and December 2019

Exclusion Criteria:

* Initial and direct preferance of open method
* Being diagnosed with malignity after histopathological evaluation
* Being operated just before one week after ERCP or after more than six weeks after ERCP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients operated with the diagnosis of acute cholecystitis a single center between January 2016 and December 2019.
Sampling Method: Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Subtotal Cholecystectomy Rate | Intraoperative
  Rate of patients needed subtotal cholecystectomy after initial intent of starting laparoscopic to the cholecystectomy

SECONDARY OUTCOMES:
Conversion to open | Intraoperative
  Rate of patients needed conversion to open after initial intent of starting laparoscopic to the cholecystectomy

OTHER OUTCOMES:
Complications | Postoperative first 90 days
  Any complications experienced by patients who underwent emergency operation with the diagnosis of acute cholecystitis
Serious complications | Postoperative first 90 days
  Any complications that has a Clavien-Dindo Score ≥ 3 experienced by patients who underwent emergency operation with the diagnosis of acute cholecystitis. (Clavien Dindo Score System that classifying post-operative complications in 5 main levels. Higher the score, the more significant complications. While level 1 is the lightest, level 5 means death)
Duration of operation | Intraoperative
  Duration of emergency with the diagnosis of acute cholecystitis
Length of hospital stay | Postoperative first 90 days
  Number of days patient stayed with and after the emergency operation with the diagnosis of acute cholecystitis
Mortality | Postoperative first 90 days
  Number of patients that died after the emergency operation with the diagnosis of acute cholecystitis

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Karabulut, Study Chair — University of Health Sciences, Bakirkoy Dr.Sadi Konuk Training and Research Hospital
Locations (1):
- Bakırkoy Dr.Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No